CLINICAL TRIAL: NCT05236803
Title: Better Understand Motor Deficits Associated With Autism Spectrum Disorders: Development of an Assessment Protocol
Acronym: MOTRICITE TSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02426-35
Record Dates: First submitted 2021-12-15; First posted 2022-02-11 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autisme Spectrum Disorders; Motricity; Cognitive disorders; Behaviour; motor skill differences
MeSH Terms: conditions — Autism Spectrum Disorder; Cognitive Dysfunction; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiology (Other): Recording of participant's performance during eye, fine motor and gross motor tests Passing self and hetero questionnaires.
  Interventions: Behavioral: Testing of general motor skills, fine motor skills and occulomotricity; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Testing of general motor skills, fine motor skills and occulomotricity — Recording of participant's performance during eye, fine motor and gross motor tests; Children's gross motor skills will be assessed through a biomechanical analysis.
  Eye movements will be recorded using the eye-tracking system (Tobii Pro TX300). The technique used is the corneal reflection technique.
Behavioral: Questionnaires — Passing self and hetero questionnaires.

SUMMARY:
This research is a case-control study aiming to characterize motor peculiarities (objective quantitative and qualitative measures) and its psycho-physiological correlates of children with ASD.

DETAILED DESCRIPTION:
The main objective is to measure jointly and in an automated and standardized manner the performance and motor patterns within the framework of tasks measuring the performance and patterns of general motor skills (postures, walking, coordination overall), fine motor skills (graphics, pointing task) and oculomotricity (visual orientation and control).

The secondary objective is to investigate the relationships between motor difficulties and cognitive and social disorders found in children with ASD.

* Compare the motor performance data in the 3 major motor domains with each other (overall, fine and oculomotor);
* Evaluate intergroup differences based on clinical characteristics (ADOS-2, ADI-R, CARS 2 scores), age, IQ, socio-communication profile score (SRS-2) and presence comorbidities (TADH, TDC).

ELIGIBILITY:
Inclusion Criteria :

All participants :

* Be between 6 and 11 years old
* Mastery of the French language
* Be affiliated with a Social Security scheme or benefit from affiliation by a third person
* Both parents (or the holder of legal authority) have read, understood and signed the study consent
* Be affiliated with social security

Participants with ASD should also verify the following inclusion criteria:

* Being diagnosed with ASD (DSM-V)

Exclusion Criteria :

All participants :

* Refusal to participate in the research on the part of the participant and / or holders of parental authority.
* Be a person benefiting from enhanced protection, namely : persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment.
* Have uncorrected visual or hearing problems
* To have concomitant psychotropic drug treatments not stabilized, initiated in the last 2 months: antipsychotics, mood stabilizers, anti-epileptics, psychostimulants, antidepressants.
* Have a motor handicap of the upper or lower limbs, fitted or not.
* Have diagnosed neurological or psychiatric disorders, present a general or metabolic pathology having a known impact on the child's motor skills (eg: Epilepsy, Tics and Gilles de la Tourette Syndrome, Intellectual Deficiency, Neuromuscular Syndrome, Metabolic Neurological Syndrome , neoplasms)
* Suspicion of low intellectual efficiency if at least one of the two subtests (Similarities or Matrices) of WISC V (retrieved from the medical file if the TSA participant) presents a result (standard score) strictly lower than 7.

Participants without ASD :

* Participant with ADHD (Attention Deficit Disorder with or without Hyperactivity) or CDD (Developmental Coordination Disorder)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Measurement performance of fine motor skills (graphics, pointing task) | At 3 month
  Jointly and in an automated and standardized manner, measure performance in the context of tasks measuring the performance and patterns of general motor skills (postures, walking, overall coordination), fine motor skills (graphics, pointing task) and oculomotricity (visual orientation and control).
Measurement performance of general motor skills with biomechanical analysis | At 3 month
  Jointly and in an automated and standardized manner, measure motor patterns in the context of tasks measuring the performance and patterns of general motor skills (postures, walking, overall coordination), fine motor skills (graphics, pointing task) and oculomotricity (visual orientation and control).
Measurement of oculomotricity with eye-tracking system (visual orientation and control) | At 3 month
  Jointly and in an automated and standardized manner, motor patterns in the context of tasks measuring the performance and patterns of general motor skills (postures, walking, overall coordination), fine motor skills (graphics, pointing task) and oculomotricity (visual orientation and control).

SECONDARY OUTCOMES:
Motor performance : success, error rate (%) | At visit 1 and visit 2, an average of 3 months
Motor performance : task duration (ms), reaction time (ms) and latency (ms) | At visit 1 and visit 2, an average of 3 months
IQ as assessed using WISC IV | At visit 1 and visit 2, an average of 3 months
Score of socio-communicative skills as assessed using Social Responsiveness Scale | At visit 1 and visit 2, an average of 3 months
  Social Responsiveness Scale :
  Min = 30, Max=90 Higher scores mean a worse outcome
ADHD as assessed using Conners-3 | At visit 1 and visit 2, an average of 3 months
Developmental Coordination Disorder as assessed using Developmental Coordination Disorder Questionnaire | At visit 1 and visit 2, an average of 3 months
  Developmental Coordination Disorder Questionnaire :
  Min = 15, Max = 75 Higher scores mean a better outcome
ASD Clinical Assessment as assessed using Childhood Autism Rating Scale | At visit 1 and visit 2, an average of 3 months
  Childhood Autism Rating Scale :
  Min = 0, Max = 100 Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Anouck AMESTOY, MD, Study Director — Physician
Locations (4):
- France (4):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Centre Hospitalier La Rochelle Re Aunis, La Rochelle
  - CHU de LIMOGES, Limoges
  - Centre Hospitalier Henri Laborit, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biffi E, Costantini C, Ceccarelli SB, Cesareo A, Marzocchi GM, Nobile M, Molteni M, Crippa A. Gait Pattern and Motor Performance During Discrete Gait Perturbation in Children With Autism Spectrum Disorders. Front Psychol. 2018 Dec 11;9:2530. doi: 10.3389/fpsyg.2018.02530. eCollection 2018. PMID 30618953
- [Result] Cazalets JR, Bestaven E, Doat E, Baudier MP, Gallot C, Amestoy A, Bouvard M, Guillaud E, Guillain I, Grech E, Van-Gils J, Fergelot P, Fraisse S, Taupiac E, Arveiler B, Lacombe D. Evaluation of Motor Skills in Children with Rubinstein-Taybi Syndrome. J Autism Dev Disord. 2017 Nov;47(11):3321-3332. doi: 10.1007/s10803-017-3259-1. PMID 28748333
- [Result] D'Mello AM, Stoodley CJ. Cerebro-cerebellar circuits in autism spectrum disorder. Front Neurosci. 2015 Nov 5;9:408. doi: 10.3389/fnins.2015.00408. eCollection 2015. PMID 26594140
- [Result] Eggleston JD, Harry JR, Cereceres PA, Olivas AN, Chavez EA, Boyle JB, Dufek JS. Lesser magnitudes of lower extremity variability during terminal swing characterizes walking patterns in children with autism. Clin Biomech (Bristol). 2020 Jun;76:105031. doi: 10.1016/j.clinbiomech.2020.105031. Epub 2020 May 7. PMID 32408186
- [Result] Hak L, Houdijk H, Beek PJ, van Dieen JH. Steps to take to enhance gait stability: the effect of stride frequency, stride length, and walking speed on local dynamic stability and margins of stability. PLoS One. 2013 Dec 13;8(12):e82842. doi: 10.1371/journal.pone.0082842. eCollection 2013. PMID 24349379